CLINICAL TRIAL: NCT00304018
Title: Pilot Study of Umbilical Cord Blood Transplantation in Adult Patients With Advanced Hematopoietic Malignancies
Brief Title: Donor Umbilical Cord Blood Transplant in Treating Patients With Advanced Hematologic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000463370; UCSF-02253; UCSF-H24045-21269-04; UCSF-2207
Record Dates: First submitted 2006-03-15; First posted 2006-03-17 (Estimated); Last update posted 2013-08-14 (Estimated); Status verified 2013-08

CONDITIONS: Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes
Keywords: adult acute myeloid leukemia with 11q23 (MLL) abnormalities; recurrent adult acute myeloid leukemia; secondary acute myeloid leukemia; adult acute myeloid leukemia in remission; adult acute erythroid leukemia (M6); adult acute megakaryoblastic leukemia (M7); adult acute monoblastic leukemia (M5a); adult acute monocytic leukemia (M5b); refractory multiple myeloma; adult acute lymphoblastic leukemia in remission; accelerated phase chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; relapsing chronic myelogenous leukemia; chronic phase chronic myelogenous leukemia; stage II multiple myeloma; stage III multiple myeloma; recurrent adult acute lymphoblastic leukemia; recurrent adult diffuse large cell lymphoma; stage III adult diffuse large cell lymphoma; recurrent mantle cell lymphoma; stage III mantle cell lymphoma; recurrent adult Hodgkin lymphoma; stage III adult Hodgkin lymphoma; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; recurrent adult T-cell leukemia/lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult Hodgkin lymphoma; stage IV adult T-cell leukemia/lymphoma; stage IV mantle cell lymphoma; stage III adult T-cell leukemia/lymphoma; stage I multiple myeloma
MeSH Terms: conditions — Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Congenital Abnormalities; Leukemia, Myeloid, Acute; Leukemia, Erythroblastic, Acute; Leukemia, Megakaryoblastic, Acute; Leukemia, Monocytic, Acute; Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Leukemia, Myeloid, Chronic-Phase; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Mantle-Cell; Hodgkin Disease; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma | interventions — Antilymphocyte Serum; sargramostim; Busulfan; Etoposide; fludarabine phosphate; Prednisone; Tacrolimus; Cord Blood Stem Cell Transplantation

ARMS (1):
- cord blood transplant (Experimental)
  Interventions: Biological: anti-thymocyte globulin; Biological: sargramostim; Drug: busulfan; Drug: etoposide; Drug: fludarabine phosphate; Drug: prednisone; Drug: tacrolimus; Procedure: allogeneic hematopoietic stem cell transplantation; Procedure: umbilical cord blood transplantation

INTERVENTIONS:
Biological: anti-thymocyte globulin
Biological: sargramostim
Drug: busulfan
Drug: etoposide
Drug: fludarabine phosphate
Drug: prednisone
Drug: tacrolimus
Procedure: allogeneic hematopoietic stem cell transplantation
Procedure: umbilical cord blood transplantation

SUMMARY:
RATIONALE: Giving chemotherapy, such as fludarabine, busulfan, and etoposide, before a donor umbilical cord blood stem cell transplant helps stop the growth of cancer cells. When the healthy stem cells from a donor are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. Sometimes the transplanted cells from a donor can make an immune response against the body's normal cells. Giving antithymocyte globulin before transplant and tacrolimus and prednisone after transplant may stop this from happening.

PURPOSE: This phase I trial is studying how well donor umbilical cord blood transplant works in treating patients with advanced hematologic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the safety and feasibility of performing donor umbilical cord blood transplantation (UCBT) in patients with advanced hematologic malignancies, in terms of > 80% engraftment rate at day 100 post-transplant and ≤ 50% transplant-related mortality.

Secondary

* Determine the toxicity of a myeloablative preparative regimen comprising busulfan, fludarabine, and etoposide prior to UCBT in these patients.
* Determine the neutrophil and platelet recovery in patients treated with this regimen.
* Determine the event-free and overall survival of patients treated with this regimen.
* Evaluate lineage-specific chimerism after UCBT and assess the contribution of each individual cord blood unit to post-transplantation hematopoiesis in these patients.
* Determine the incidence, severity, and timing of acute and chronic graft-vs-host disease in patients treated with this regimen.

OUTLINE: This is a pilot study.

* Preparative regimen: Patients receive fludarabine IV over 30 minutes on days -7 to -3, busulfan IV over 2 hours 4 times daily on days -7 and -4, etoposide IV over 4 hours on day -3, and anti-thymocyte globulin IV over 6 hours on days -2 and -1.
* Donor umbilical cord blood transplantation (UCBT): Patients undergo donor UCBT on day 0. Beginning on day 7, patients receive sargramostim (GM-CSF) IV or subcutaneously once daily until blood counts recover.
* Graft-vs-host disease prophylaxis: Patients receive tacrolimus IV continuously over 24 hours or orally twice daily beginning on day -2 and continuing until day 180 followed by a taper. Patients also receive oral prednisone twice daily on days 13-50 and then once daily on days 50-60, followed by a rapid taper.

After completion of study treatment, patients are followed periodically for approximately 2 years.

PROJECTED ACCRUAL: A total of 10 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of 1 of the following advanced hematologic malignancies:

  * Acute myeloid leukemia (AML) meeting the following criteria:

    * Not expected to be curable with chemotherapy and meets ≥ 1 of the following criteria:

      * High-risk cytogenetics (-7, -7q, -5, -5q, t[6,9], t[9,11], complex, Philadelphia chromosome positive [Ph+])
      * AML evolved from prior myelodysplasia
      * AML secondary to prior chemotherapy
      * Failed to achieve remission
      * In second or subsequent remission
    * Marrow blasts ≤ 10% (may be achieved using chemotherapy)
  * Myelodysplastic syndromes (MDS) with high-risk features

    * International Prognostic Scoring System (IPSS) score intermediate -2 or high-risk
    * Marrow blasts ≤ 20% (may be achieved using chemotherapy)
  * Acute lymphoblastic leukemia meeting the following criteria:

    * Not expected to be curable with chemotherapy and meets ≥ 1 of the following criteria:

      * High-risk cytogenetics (Ph+, t[4,11], 11q23 abnormalities, and monosomy 7)
      * Required > 1 induction course to achieve remission
      * Failed to achieve remission
      * In second or subsequent remission
    * Marrow blasts ≤ 10% (may be achieved using chemotherapy)
  * Chronic myelogenous leukemia meeting ≥ 1 of the following criteria:

    * Accelerated phase
    * Chronic phase refractory to imatinib mesylate
    * Blastic phase

      * Marrow blasts ≤ 10% (may be achieved using chemotherapy)
  * Multiple myeloma meeting 1 of the following criteria:

    * Stage II or III disease with > first relapse or refractory disease
    * Newly diagnosed disease with chromosome 13 abnormalities
  * Lymphoma meeting the following criteria:

    * One of the following subtypes:

      * Diffuse large cell lymphoma
      * Mantle cell lymphoma
      * Peripheral T-cell lymphoma
      * T-natural killer (NK) cell lymphoma
      * Hodgkin's lymphoma
    * Disease failed to respond to primary therapy, progressed, or recurred after prior therapy

      * Patients who have failed autologous stem cell transplantation are eligible provided it has been > 1 year since transplant
* No rapid progression of malignant disease
* Not eligible for autologous stem cell transplantation
* Available umbilical cord blood (1-3 units) donor matching at ≥ 4 of 6 HLA antigens (A, B, and DR)

  * Patients with an HLA-identical or 1 antigen-mismatched related donor OR a potential HLA-matched unrelated donor matching at > 6/8 (A, B, C, DR) alleles are not eligible

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Creatinine < 2.0 mg/dL
* Creatinine clearance > 40 mL/min
* Bilirubin < 2.0 mg/dL
* AST and alkaline phosphatase < 3 times upper limit of normal
* Hepatitis C and active hepatitis B allowed if patient has ≤ grade 2 inflammation or fibrosis by liver biopsy
* Ejection fraction > 40% by echocardiogram or MUGA
* DLCO > 40% of predicted
* Not pregnant or nursing
* Negative pregnancy test
* No known HIV infection
* No active infection requiring ongoing antibiotic treatment

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2002-10; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Determine the safety and feasibility of performing donor umbilical cord blood transplantation (UCBT) in patients with advanced hematologic malignancies | up to 24 months post-transplant
  Determine the safety and feasibility of performing donor umbilical cord blood transplantation (UCBT) in patients with advanced hematologic malignancies, in terms of > 80% engraftment rate at day 100 post-transplant and ≤ 50% transplant-related mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas G. Martin, MD, Study Chair — University of California, San Francisco
Locations (1):
- UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California, United States